CLINICAL TRIAL: NCT00795210
Title: Effects of Short-term Growth Hormone in HIV-infected Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Steven K. Grinspoon, MD, Professor of Medicine, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DK63639A; R01DK063639 (NIH)
Record Dates: First submitted 2008-11-20; First posted 2008-11-21 (Estimated); Results first posted 2014-01-08 (Estimated); Last update posted 2014-01-08 (Estimated); Status verified 2013-10

CONDITIONS: HIV Lipodystrophy
Keywords: HIV lipodystrophy; growth hormone; growth hormone releasing hormone
MeSH Terms: interventions — Growth Hormone; Growth Hormone-Releasing Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- GH 6mcg/kg/d (Experimental): Recombinant human growth hormone 6mcg/kg SC once daily
  Interventions: Drug: Growth hormone
- GH 2mg daily (Experimental): Recombinant human growth hormone 2mg SC once daily
  Interventions: Drug: Growth hormone
- Growth Hormone Releasing Hormone (Experimental): Growth Hormone Releasing Hormone (Tesamorelin) 2mg daily, injected subcutaneously, x 2 weeks
  Interventions: Drug: Growth Hormone Releasing Hormone

INTERVENTIONS:
Drug: Growth hormone — Recombinant Human Growth Hormone (Teva pharmaceuticals), with one arm receiving 6mcg/kg SC once daily for two weeks and the other arm receiving 2mg SC once daily for two weeks
  Other Names: rhGH from Teva Pharmaceuticals
  Arms: GH 2mg daily; GH 6mcg/kg/d
Drug: Growth Hormone Releasing Hormone — Tesamorelin (GHRH) 2mg SC QD x 2 weeks
  Arms: Growth Hormone Releasing Hormone

SUMMARY:
The purpose of this study is to examine the short-term effects of two different doses of growth hormone, compared to treatment with growth hormone releasing hormone, on the brain's secretion of growth hormone and the body's glucose metabolism. We hypothesize that growth hormone administration will alter the body's endogenous pulsatile growth hormone secretion and that higher dose growth hormone may decrease insulin sensitivity. We hypothesize that growth hormone releasing hormone will augment endogenous GH pulsatility and be neutral to insulin sensitivity.

DETAILED DESCRIPTION:
The primary objective of this study is to determine the differential effects of growth hormone releasing hormone (GHRH) vs. low dose physiologic growth hormone (GH) vs. higher dose GH treatment and withdrawal on endogenous overnight growth hormone secretion and pulsatility, as well as insulin-stimulated glucose uptake. Subjects with HIV-infection will be randomized to receive one of three treatments: GHRH 2mg/day, or growth hormone 6mcg/kg/day (physiologic "low" dose), or growth hormone 2mg/day ("higher" dose) for 2 weeks. At baseline and after two weeks of treatment, we will assess overnight growth hormone by frequent sampling as well as insulin stimulated glucose uptake by clamp. Subjects will then stop the treatment and will return for an identical assessment after a 2 week withdrawal period.

ELIGIBILITY:
Inclusion Criteria:

* previously diagnosed HIV infection
* Stable antiretroviral regimen for at least 12 weeks prior to enrollment
* Waist circumference >/= 95cm and waist-to-hip ratio >/= 0.94 for males or waist circumference >/=94cm and WHR >/= 0.88 for females, occurring in the context of treatment for HIV disease
* Subjective evidence of at least one of the following changes, occurring during the treatment of HIV disease: increased abdominal girth, relative loss of fat in the extremities, or relative loss of fat in the face

Exclusion Criteria:

* Use of anti-diabetic agents, Megace, testosterone, or any steroid use within 6 months of the study
* Use of GH or Growth hormone releasing factor within six months of starting the study
* Change in lipid lowering or antihypertensive regimen within 3 months of screening
* Fasting blood sugar >126mg/dL, SGOT > 2.5 times ULN, Hgb < 12.0 g/dL, creatinine > 1.4 mg/dL, FSH > 20 IU/L in women, or CD4 count < 200
* Carpal tunnel syndrome
* Severe chronic illness or active malignancy or history of pituitary malignancy or history of colon cancer
* For men, history of prostate cancer or evidence of prostate malignancy by PSA > 5ng/mL
* Prior history of hypopituitarism, head irradiation, or any other condition known to affect the GH axis
* positive beta-HCG (women only)
* Oral contraceptives, depo provera, or combined progesterone-estrogen injections, transdermal contraceptive patches, estrogen or progestin coated IUD's within 6 months of the study
* weight < 110 pounds

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2009-02; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven K Grinspoon, M.D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- MGH, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred between January, 2009 and November, 2012, in the Boston area.
Pre-assignment Details: Once patients were found to be eligible (after screen visit) and agreed to participate, there were no additional events prior to baseline.
Period: Overall Study
Arm/Group | GH 6mcg/kg/d | GH 2mg Daily | Growth Hormone Releasing Hormone
Started | 8 | 12 | 5
Completed | 8 | 11 | 3
Not Completed | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GH 6mcg/kg/d | GH 2mg Daily | Growth Hormone Releasing Hormone | Total
Number analyzed (Participants) | 8 | 12 | 5 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 12 | 5 | 25
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 49 (7) | 49 (6) | 47 (4) | 48 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 0 | 2
  Male | 8 | 10 | 5 | 23
Region of Enrollment [Number; unit: participants]
  United States | 8 | 12 | 5 | 25

OUTCOME MEASURES:

1. Primary Outcome: Overnight Mean Growth Hormone Secretion After 2 Weeks of Study Drug
Description: Serum was sampled for growth hormone concentrations every 20 minutes between 20:00 (8pm) and 07:40 (7:40am). Subjects in GH 6mcg/kg/day and GH 2mg daily groups received their final dose of study drug approximately 36 hours prior to start of sampling. Subjects in Growth Hormone Releasing Hormone group received their final dose of study drug approximately 8 hours prior to start of sampling.
Time Frame: after 2 weeks treatment
Population: Overnight GH data were unavailable for 1 subject in the GH 6mcg/kg group and thus are not included in analysis.
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | GH 6mcg/kg/d | GH 2mg Daily | Growth Hormone Releasing Hormone
Number analyzed (Participants) | 7 | 11 | 3
ng/mL | 0.23 [0.08 to 0.68] | 0.07 [0.04 to 0.12] | 1.24 [0.76 to 1.52]
Statistical Analysis 1: Comparison: GH 6mcg/kg/d vs GH 2mg Daily vs Growth Hormone Releasing Hormone; Kruskal-Wallis Test for overall difference between groups; Test type: Superiority or Other; p = 0.01, Kruskal-Wallis

2. Secondary Outcome: Insulin Sensitivity
Description: insulin-stimulated glucose uptake as measured by euglycemic hyperinsulinemic clamp; "M" value (infusion rate with space correction, using method of DeFronzo) for the steady state between 100-120 minutes of clamp is given
Time Frame: after two weeks treatment
Population: Insulin stimulated glucose uptake data were unavailable for 4 subjects in the GH 2mg group. Two subjects did not have sufficient IV access and thus could not complete the clamp procedure. Two subjects did not reach target glucose and thus their data could not be used.
Measure: Mean (Standard Deviation); unit: mg/kg/min
Arm/Group | GH 6mcg/kg/d | GH 2mg Daily | Growth Hormone Releasing Hormone
Number analyzed (Participants) | 8 | 7 | 3
mg/kg/min | 9.0 (2.9) | 7.5 (3.2) | 9.9 (1.2)
Statistical Analysis 1: Comparison: GH 6mcg/kg/d vs GH 2mg Daily vs Growth Hormone Releasing Hormone; Test type: Superiority or Other; p = 0.42, ANOVA

ADVERSE EVENTS:
Time Frame: AE data were actively collected during the 4 weeks of the study period.
Arm/Group | GH 6mcg/kg/d | GH 2mg Daily | Growth Hormone Releasing Hormone
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/11 | 0/3
Other Adverse Events (participants affected / at risk) | 1/8 | 3/11 | 2/3
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GH 6mcg/kg/d (N=8) | GH 2mg Daily (N=11) | Growth Hormone Releasing Hormone (N=3)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Sinus Infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Edema/Extremity Swelling (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0)
hyperglycemia (Endocrine disorders) | 0 (0) | 2 (2) | 0 (0) — elevated fasting blood sugar
injection site bruising (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The study was completed early due to the lack of availability of study drug for one of the arms.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No